CLINICAL TRIAL: NCT05510674
Title: Safety and Dose Ranging Study for OWL-EVO1 as a Lung Cancer EVOC® Probe
Brief Title: Safety and Dose Ranging Study for OWL-EVO1 as a Lung Cancer EVOC® Probe (Evolution)
Acronym: Evolution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Owlstone Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OML-001
Record Dates: First submitted 2022-04-04; First posted 2022-08-22 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Diagnostic Test; Diagnostic Breath Test
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OWL-EVO1 (Experimental): OWL-EVO1 probe will be administered to those who are fully eligible, including those diagnosed with lung cancer and healthy volunteers
  Interventions: Diagnostic Test: OWL-EVO1

INTERVENTIONS:
Diagnostic Test: OWL-EVO1 — EVOC probe
  Other Names: OWL-EVO1 Breath Biopsy Test; D5-ethyl-βD-glucuronide

SUMMARY:
The Evolution study is a phase 1a and 1b study evaluating the safety and pharmacokinetics of D5- ethyl-βGlucuronide as well as the target dose for the probe to maximize the difference between controls and subjects with lung cancer.

The phase 1a study will be designed as a single ascending dose study in healthy volunteers and will be conducted in a phase 1 trial unit with a primary objective to assess safety of the probe. A subsequent phase 1b study will be conducted at clinical sites and will aim to find the optimal dosing and breath sampling protocol to maximize the accuracy of the breath test.

Evolution Phase 1 is a multicentre study; Phase 1a will be conducted at a Phase 1 facility in Belgium and Phase 1b will be conducted in the UK.

DETAILED DESCRIPTION:
Owlstone has recently pioneered the EVOC approach which enables active investigation of disease specific pathways by administering probe compounds to patients and measure its signal on breath. In the Evolution study, Owlstone Medical aims to evaluate one such EVOC probe strategy based on the administration of the probe OWL-EVO1.

The Evolution study consist of phase 1a, in which the safety and pharmacokinetics of OWL-EVO1 are assessed; in this part of the study up to 21 healthy volunteers will be recruited. The probe will be administered for the first time in humans in a single ascending dose design. Five different doses of the probe are planned to be administered across 5 different cohorts. This part of the study will be conducted at a Phase 1 unit in Belgium. Participating subjects will be administered a dose of the EVOC probe; up to 8 breath samples, using Owlstone's RECIVA, will be collected in a 24h wash-out.

In the subsequent Phase 1b, research will aim to identify the most optimal dose and timing of the breath test to maximise the discriminative signal between lung cancer patients (cases) and healthy controls. Up to 50 cases and 50 controls will be recruited in selected sites in the UK. The Phase 1b has been designed as an adaptive trial design. Participating subjects will be administered the probe and will provide up to 7 breath samples over a 240 minute wash-out.

This study is intended to provide proof of concept for the use of OWL-EVO1 as a probe for breath-based detection of lung cancer.

This will be an important step towards creating a breath-based screening approach for lung cancer.

ELIGIBILITY:
Inclusion Criteria:Phase 1a

1. Aged 18-70 years
2. Ability to provide written informed consent
3. Weight not exceeding 100 kg
4. Body Mass Index (BMI) between 18.5 and 30
5. Meeting criteria for fitness for infusion as detailed in Section 10.3.1 - Safety Assessment Phase 1a and b Study

Inclusion Criteria: Phase 1b

1. Aged 55-80 years
2. Ability to provide informed consent
3. Weight not exceeding 100kg
4. BMI between 18.5 and 30.0
5. Meeting criteria for fitness for infusion as detailed in Section 10.3.1 - Safety Assessment Phase 1a and b Study

Control specific inclusion criteria - phase 1b ONLY 1. healthy as per medical records and clinical assessment at screening

Lung cancer subject specific inclusion criteria - Phase 1b ONLY

1. Tumor Node Metastasis (TNM) stage I, II, III or IV primary lung cancer.
2. Multi-Disciplinary Team (MDT) diagnosis of an invasive malignant lung tumor. This evaluation should integrate data from the clinical, imaging and pathology work-up.

Exclusion Criteria:

Phase 1a and 1b

1. (Anticipated) inability to complete the breath sampling procedure due to e.g., inability to maintain adequate ventilation unaided or claustrophobia.
2. Received an investigational medical product in the context of a Clinical Trial (CTIMP)during the 28 days prior to first probe administration.
3. History of alcohol dependence or diagnosis of alcoholism.
4. Subjects known to suffer from an unstable systemic, inflammatory, infectious, or neoplastic condition. Specifically, subjects should be excluded if:

   4.1. Currently in the process of investigation for a potential malignancy. 4.2. Any history of cancer or indeterminate lung nodule. 4.3. Known active bacterial, fungal, or viral infection including but not limited to upper respiratory tract infection, tuberculosis, pneumonia, cystitis, pyelonephritis, active gastritis under medical treatment, prostatitis, or viral hepatitis. Patients can be recruited after being symptom free for at least 2 weeks for mild infections or 6 weeks if admitted to the hospital and/or treated with intravenous antibiotics. For the avoidance of doubt: Any skin infection without subcutaneous involvement (such as acne vulgaris) is permissible in the study.

   4.4. Clinically diagnosed presence of rheumatoid arthritis. Osteoarthritis, spondylarthritis and sports injuries are NOT exclusion criteria 28.

   4.5. Documented history of a clinically important lung condition including asthma, Chronic Obstructive Pulmonary Disease (COPD), α1- antitrypsin deficiency, moderate to severe bronchiectasis and/or exacerbation of bronchiectasis requiring treatment, cystic fibrosis, primary ciliary dyskinesia, allergic bronchopulmonary aspergillosis/mycosis, moderate to severe pulmonary fibrosis or hypersensitivity pneumonitis.

   4.6. Known renal function impairment (eGFR 45ml/min or less). 4.7. Known liver function impairment with test results being above 1.5 times the normal upper limit.

   4.8. Pregnant or breastfeeding women and women of child-bearing potential not using adequate contraceptive methods. Please refer to Appendix 1 for an overview of highly effective contraceptive measures that are accepted adequate contraceptive methods for this study. A woman of childbearing potential is a woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient any hospitalization during the 6 weeks prior to first probe administration.
5. Known glucose intolerance or Diabetes Mellitus.
6. Self-reported immunocompromised patients: specifically, patients with Acquired Immune Deficiency Syndrome (AIDS), inborn or acquired severe immunodeficiency including those caused by pharmacological treatment.
7. Documented history of pulmonary surgery or endobronchial interventional procedures other than biopsy, lavage, or bronchial brushings. These include surgical resection,

Control specific exclusion criteria - phase 1b ONLY

1. Under clinical investigation for lung cancer
2. Current smoker
3. At high risk of lung cancer: Aged 55-70 with >30 packyears smoking history, either a current smoker or quit smoking in the past 15 years as per USPSTF risk-criteria30.

Lung cancer subject specific exclusion criteria - phase 1b ONLY

1. Initiation of treatment for lung cancer prior to providing final breath sample.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Confirm safety of OWL-EVO1 probe in Phase 1a | 2 months
  The primary endpoint for the Phase 1a study is safety of OWL-EVO1 being administered to the subjects evaluated through the number of adverse events and whether or not they are related to the administered probe.
Determining optimal dose | 8 months
  To determine the optimal dose(mg/kg) of the OWL- EVO1 breath test which maximizes the discriminative signal between cases and controls
Evaluate the safety safety of OWL-EVO1 probe in Lung cancer patients | 8 months
  The primary endpoint for the Phase 1b study is to evaluate safety of OWL-EVO1 in healthy subjects and Lung cancer patients.
Determining optimal timing | 8 months
  To determine the optimal timing (minutes) of the OWL- EVO1 breath test which maximizes the discriminative signal between cases and controls

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rintoul, Principal Investigator — Royal Papworth Hospital
Locations (2):
- United Kingdom (2):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire
  - Wythenshawe Hospital, Manchester, Greater Manchester

IPD SHARING:
Plan to Share IPD: No